CLINICAL TRIAL: NCT01975974
Title: Technique for Successful Ultrasound-guided Peripheral Vascular Access
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Kenichi Ueda, Clinical Associate Professor, University of Iowa
Other Study IDs: 201307701
Record Dates: First submitted 2013-08-02; First posted 2013-11-05 (Estimated); Results first posted 2016-12-20 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Obesity; Vascular Diseases
Keywords: vascular; access; ultrasound
MeSH Terms: conditions — Obesity; Vascular Diseases | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ultrasound: Ultrasound guided peripheral vascular access
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Using ultrasound as a guide for peripheral venous cannulation in obese patients

SUMMARY:
Obtaining peripheral vascular access in medical patients is a necessary procedure for many healthcare providers. Peripheral vascular access is traditionally performed using palpation or visual inspection to identify appropriate points of entry in the vasculature after which a needle and catheter are threaded through the skin and surround fascia into the vessel of interest. This procedure, one of the most common procedures in the medical field including both artery and vein access, is not 100% successfully attempted. Operator skill heavily influences peripheral vascular cannulation. (Frisch et al. 2013) However, certain patient populations have difficult peripheral vessels to identify by palpation or visual inspection and past operators would be forced to perform the procedure blind based on anatomical landmarks. Recently, to aid vascular identification and increase cannulation success, a number of alternative techniques for peripheral vascular access have been described including ultrasound-guided.

Ultrasound-guided vascular access has been utilized in vascular access with improved success rate. However, even with ultrasound guidance the first attempt success rate of cannulation was only approximately 65%. A proposed failure of ultrasound guided peripheral vascular access is most likely due to failure to advance the catheter into the vessel even the vessel was successfully punctured. The investigators propose a specific technique and the positive "Target Sign" as a means to obtain almost 100% successful peripheral vascular access.

The investigators plan to enroll 100 surgical patients in the above study and study procedures will not differ from what a patient in the operating room under the care of anesthesia faculty would receive. The above study is simply a way to identify the steps regarding a specific technique.

DETAILED DESCRIPTION:
The subjects (patients) will be brought to the Main Operating Room after their time in the Day of Surgery Admissions (DOSA) at the discretion of the attending physicians and surgical team. The patients will not be required to do anything different from standard anesthesia and surgical practice at the hospital. Subjects will come to the operating room suite and the usual monitors (electrocardiogram, non-invasive blood pressure, and oxygen saturation) will be placed.

Prior to the routine induction of anesthesia, peripheral vascular access is usually obtained. In regards to the subject population, peripheral vascular access is predicted to be more difficult due to lack of visualization of the peripheral vessels. The skin will be prepped with chlorhexidine, draped, and all subsequent procedures will be performed in sterile fashion. The attending physician and/or resident will use the L25x Sonosite transducer with the Sonosite Edge® (Washington, US) to identify a peripheral vessel in the upper extremity for cannulation. After identification of the vessel, the operator will line the L25x Sonosite transducer to place the vessel horizontally midline on the Sonosite Edge® screen to give the most available viewing area. A BD Insyte® Autoguard® 16G shielded IV catheter (Becton Dickinson Infusion Therapy Systems Inc., Utah, US) will be advanced toward the vessel at an approximately 10˚ angle. Once the needle tip is identified on the Sonosite Edge® monitor in short axis view, the following steps will ensue:

1. Advance the needle toward the vessel slowly, adjusting the ultrasound transducer position and angle to continue to keep the needle tip and vessel identified on the Sonosite Edge® monitor.
2. Puncture the anterior wall of the vessel with the needle tip
3. Confirm needle tip placement in vessel
4. Advance the needle within the vessel 5mm under continuous visualization
5. View and record confirmation of "Target Sign" on ultrasound monitor

   1. Positive Target Sign=needle tip is identified on ultrasound monitor within vessel and is able to move freely within the vessel, similar to a circle with a target in the middle which is able to move. This confirms the needle is unrestricted in the vessel.
   2. Negative Target Sign=needle is identified on ultrasound monitor within vessel, but is unable to move freely within the vessel without dragging the vessel wall with needle movement. This confirms the needle is transfixed on the posterior wall of the vessel
6. Thread the catheter over the needle.
7. At this point, the catheter could be advanced either with or without a guidewire at the operator's discretion Members of the research team will be available for verbal assistance throughout this procedure.

Number of attempts and time to successful vessel cannulation will be measured, starting from when either the operator's fingers or the ultrasound probe made contact with the patient's skin. Successful vessel cannulation will be defined as a flowing IV bag of saline after connection and confirmation of flow via fluid agitation in vessel identified via ultrasound.

This procedure will be incorporated in the subjects standard of care and will not extend the time of operation.

At this point, patient participation in the study will be over and surgical operation under the discretion of the surgical team. The video recording of the Target Sign will be saved and given to a member of the research team unknowing of the success of the cannulation. The member of the research team will decide, based on the ultrasound video recording of a positive or negative Target Sign, if the cannulation was successful or unsuccessful. The viewer will record his/her answers and compare with the actual result of the cannulation.

Analysis of unsuccessful and successful cannulations will be compared with a Positive or Negative Target Sign. No additional long-term followup will occur.

ELIGIBILITY:
Inclusion Criteria:

1. morbid obese surgical patients requiring large bore IV.
2. no visible intravenous access in upper arm

Exclusion Criteria:

1) No target vein by US screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be surgical patients requiring peripheral intravenous access.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Ueda, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hosptials and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
we are not planning on sharing the data

REFERENCES:
- [Derived] Ueda K, Hussey P. Dynamic Ultrasound-Guided Short-Axis Needle Tip Navigation Technique for Facilitating Cannulation of Peripheral Veins in Obese Patients. Anesth Analg. 2017 Mar;124(3):831-833. doi: 10.1213/ANE.0000000000001653. PMID 27984247

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasound
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ultrasound
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 54

OUTCOME MEASURES:

1. Primary Outcome: Successful First Attempt Peripheral Venous Cannulation
Description: we will compare the first attempt success rate using proposed ultrasound technique in total of 100 obese (BMI>30) surgical patients with existing published data. Mata-analysis of first attempt success rate using ultrasound for intravenous cannulation is 61.8% We predict 90% (50% improvement) success rate using the proposed ultrasound technique. Based on this prediction, a sample size of 100 patients provided more than 90% power to compare there two groups at the 0.05 significance level with a two-sided Chi square test.
Time Frame: one day
Measure: Number; unit: participants
Arm/Group | Ultrasound
Number analyzed (Participants) | 100
participants | 96

ADVERSE EVENTS:
Arm/Group | Ultrasound
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 1/100
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrasound (N=100)
IV infiltration (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No